CLINICAL TRIAL: NCT07218328
Title: Food is Medicine in Survivorship: Examining the Feasibility and Impact of a Scalable Food Delivery and Culinary Medicine Program (FoodiiS) Among Pediatric Cancer Survivors and Their Families
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2025-1327; NCI-2025-07664 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-10-16; First posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Pediatric Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Waitlist Control (No Treatment until after T1 and then Access to all FoodiiS Materials) (Experimental): Target participants for this study will be parents/guardians of school-aged (5-12 years) pediatric cancer survivors that are within first 5 years off active treatment.
  Interventions: Dietary Supplement: FoodiiS plus Culinary Essentials Food Delivery; Dietary Supplement: Waitlist control
- FoodiiS (Digital Culnary Medicine Intervention + Culinary Essentials Food Delivery) (Experimental): Target participants for this study will be parents/guardians of school-aged (5-12 years) pediatric cancer survivors that are within first 5 years off active treatment.
  Interventions: Dietary Supplement: Culinary Essentials Food Delivery Only
- Culinary Essential Food Delivery Alone (No Other Intervention) (Experimental): Target participants for this study will be parents/guardians of school-aged (5-12 years) pediatric cancer survivors that are within first 5 years off active treatment.
  Interventions: Dietary Supplement: Waitlist control

INTERVENTIONS:
Dietary Supplement: FoodiiS plus Culinary Essentials Food Delivery — The FoodiiS intervention will include videos, recipes, and other online healthy eating content adapted from previously developed materials.
  Arms: Waitlist Control (No Treatment until after T1 and then Access to all FoodiiS Materials)
Dietary Supplement: Culinary Essentials Food Delivery Only — To support participants in effectively learning the healthy cooking strategies and mitigate access issues, investigators will provide participating families two home food deliveries of non-perishable culinary ingredients that are related to HCI practices including whole grain versions of common products (brown rice, whole wheat flour), healthier cooking oils (olive and canola), and a core selection of herbs and spices, among other goods.
  Arms: FoodiiS (Digital Culnary Medicine Intervention + Culinary Essentials Food Delivery)
Dietary Supplement: Waitlist control — The control group will receive no intervention until after T1. After the T1 data collection time point, the control group will receive all FoodiiS intervention materials.
  Arms: Culinary Essential Food Delivery Alone (No Other Intervention); Waitlist Control (No Treatment until after T1 and then Access to all FoodiiS Materials)

SUMMARY:
The goal of this research study is to learn if the FoodiiS-Kids intervention is useful to parents and guardians of pediatric cancer survivors.

DETAILED DESCRIPTION:
Primary Objective:

Assess the feasibility and acceptability of the FoodiiS intervention for parents of pediatric cancer survivors (recruitment, retention, satisfaction).

Secondary Objective:

Explore the preliminary efficacy of FoodiiS to improve diet quality and cooking behaviors among parents of pediatric cancer survivor.

ELIGIBILITY:
Inclusion Criteria:

* Parents/guardians of school-aged (5-12 years) pediatric cancer survivors.
* Have children that are within five years of having completed active treatment.
* Self-report having internet access.
* Self-report as being able to speak and read English.
* Willing to complete study assessments.

Exclusion Criteria:

* Parents of pediatric cancer survivors over 12 years of age.
* Unwilling or unable to complete study assessments.
* Self-report to not speak English.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2026-04-30 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Marget Raber, DRPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org